CLINICAL TRIAL: NCT02370979
Title: Impact of Starting a Dolutegravir-based Regimen on HIV-1 Proviral DNA Reservoir Of Treatment Naïve and Experienced Patients
Acronym: DRONE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5973
Record Dates: First submitted 2015-01-26; First posted 2015-02-25 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: HIV-1 Infection
Keywords: Dolutegravir; Proviral HIV-1 DNA; Reservoir
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dolutegravir (Experimental)
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples

SUMMARY:
This is a multi-center prospective study. The primary objective of DRONE study is to investigate the change of the size of HIV-1 DNA reservoir in blood from baseline to week 48 (W48) in participants treated by DTG-based regimen. Secondary objectives include: DTG pharmacokinetic and analysis of biomarkers of immune activation from baseline to W48.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged from de 18 to 80 years
* Patient starting a DTG-regimen
* Patients agreeing to use methods of birthcontrol while on the study and during the 6 weeks after stopping DTG treatment
* Signed and dated written informed consent is obtained from the subject or the subject's legal representative prior to screening

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* HBV or HCV coinfection
* Participation in another clinical drug or device trial where the last dose of drug was within the past 30 days or an investigational medical device is currently implanted
* An active AIDS-defining condition at Screening
* Documented resistance to DTG
* Allergy or intolerance to the study drugs or their components or drugs of their class
* Any acute or verified Grade 4 laboratory abnormality (with the exception of Grade 4 lipids) at Screening.
* Coadministration with Dofelitide

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Proviral HIV-1 DNA at Week 48 | baseline (Day 0) and Week 48

SECONDARY OUTCOMES:
Dolutegravir pharmacokinetic (dolutegravir pharmacological blood levels) | Week 4, Week 24 and Week 48
Quantification of biomarkers of immune activation | baseline (Day 0), Week 24 and Week 48
  CRPus, IL-6, neopterin, D-dimer, CD14s

CONTACTS AND LOCATIONS:
Overall Officials: David REY, PhD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (4):
- France (4):
  - Centre hospitalier de Belfort-Montbéliard, Belfort
  - Centre hospitalier de Colmar, Colmar
  - Centre hospitalier de Mulhouse, Mulhouse
  - Hôpitaux Universitaire de Strasbourg, Strasbourg